CLINICAL TRIAL: NCT04721392
Title: Mental Fatigue and Industrial Work Performance: The Influence of the Laevo Exoskeleton
Brief Title: Mental Fatigue and Industrial Work Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Prof. Dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MF-Industrial Work
Record Dates: First submitted 2020-09-22; First posted 2021-01-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Healthy; Mental Fatigue; Industrial Work; Robotics
MeSH Terms: conditions — Mental Fatigue | interventions — Stroop Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mental fatigue - No Robot (Experimental): During a 15 minute trial, the participant will relocate a box of 5 kilograms between ground level and shoulder height. During this task, the participants are asked to perform the serial seven task, continuously subtracting seven from a given number between 900 and 950. Afterwards, the participant will perform a 60- minute Stroop task and is asked to repeat this abovementioned physical dual-task.
  Interventions: Other: Mental fatigue (Stroop task)
- Mental fatigue - Exoskeleton (Experimental): During a 15 minute trial, the participant will wear the Laevo exoskeleton and will relocate a box of 5 kilograms between ground level and shoulder height. During this task, the participants are asked to perform the serial seven task, continuously subtracting seven from a given number between 900 and 950. Afterwards, the participant will perform a 60- minute Stroop task and is asked to repeat this abovementioned physical dual-task.
  Interventions: Other: Mental fatigue (Stroop task)
- No Mental fatigue - No Robot (Placebo Comparator): During a 15 minute trial, the participant will relocate a box of 5 kilograms between ground level and shoulder height. During this task, the participants are asked to perform the serial seven task, continuously subtracting seven from a given number between 900 and 950. Afterwards, the participant will watch a 60- minute neutral documentary and is asked to repeat this abovementioned physical dual-task.
  Interventions: Other: Control (documentary)
- No Mental fatigue - Exoskeleton (Placebo Comparator): During a 15 minute trial, the participant will wear the Laevo exoskeleton and will relocate a box of 5 kilograms between ground level and shoulder height. During this task, the participants are asked to perform the serial seven task, continuously subtracting seven from a given number between 900 and 950. Afterwards, the participant will watch a 60- minute neutral documentary and is asked to repeat this abovementioned physical dual-task.
  Interventions: Other: Control (documentary)

INTERVENTIONS:
Other: Mental fatigue (Stroop task) — A modified Stroop task of approximately 60 min will be used in order to induce mental fatigue (MF). This will be based on their performance during the max test that was conducted during the familiarization session. In this task, which will be partitioned in 4 blocks of 468 stimuli, four colored words ("rood", "blauw", "groen" and "geel") will be presented one at a time on a computer screen. The participants will be required to indicate the color of the word, ignoring the meaning of the word itself.
  Arms: Mental fatigue - Exoskeleton; Mental fatigue - No Robot
Other: Control (documentary) — In the control task subjects will have to watch a documentary of 60 min on the same computer screen as the one used for the experimental trial. In order to avoid under- and over-arousal the subjects will have the opportunity to choose between several documentaries as proposed by the research team.
  Arms: No Mental fatigue - Exoskeleton; No Mental fatigue - No Robot

SUMMARY:
To investigate the effect of mental fatigue on industrial work performance, biomechanical determinants, (electro-)(psycho-) physiological measures and physical ergonomics. Additionally, the current project wants to evaluate whether or not the Laevo exoskeleton influences the aforementioned parameters when mental fatigue is acutely induced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Males and Females
* 18-64 years

Exclusion Criteria:

* Musculoskeletal disorders
* Neurological disorders
* Cardiovascular disorders
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
VICON: Placement accuracy Box | 30 minutes
  Accuracy of placement box during the dual-task will be measured with VICON. VICON-markers will be placed on the box to track its movement during the trial. First, the optimal position of the box for each level (ground or shoulder) will be determined, these will form the reference frames. Next, the accuracy of each relocation will be determined by the offset compared to these reference frames. This will be calculated into a percentage.
Work performance: Percent accuracy Serial Seven Task | 30 minutes
  An audio record of this task will be made to verify made errors posthoc. During the serial seven task participants are given a number between 900 and 950. The given starting number will change each trial. Participants are asked to subsequently subtract seven as fast as possible.The researcher will take note of every answer. If the participant makes an error, he/she may continue to calculate with the wrong number. The ratio of correct answers to the total number of responses will indicate the percent accuracy for each participant.
Ergonomics: EMG-data | 30 minutes
  Muscle activity during the performance of the industrial task of the erector spinae muscle, m. rectus abdominus, both m. obliqui abdominus, all three parts of m. trapezius, all three of m. deltoideus, m. pectoralis major, m. latissimus dorsi, m. biceps brachii, m. triceps brachii,m. flexor- and extensor carpi radials, m. flexor- and extensor carpi ulnaris, m. flexor- and extensor digitorum, m. gluteus maximus and medius, m. rectus femoris, m. biceps femoris. ; measured with Cometa mini wave.
Ergonomics: Joint angles | 30 minutes
  Joint angles will be measured during the performance of the industrial task to evaluate movement variability. 30 VICON markers will be placed bilateral on the body of the participant on anatomical landmarks.
Mental fatigue: EEG-data | 60 minutes
  Alpha, Beta and Theta activity in the electroencephalogram measured with open bci (OpenBci, inc)
Mental fatigue: VAS-score | 60 minutes
  Participants are asked to indicate their subjective feeling on a straight line ranging from "not at all mentally fatigued" to "extreme mentally fatigued"

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Etterbeek, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No